CLINICAL TRIAL: NCT07267078
Title: Neoadjuvant Tuvonralimab and Iparomlimab With Gemcitabine-oxaliplatin for Biliary Tract Cancer
Brief Title: Tuvonralimab and Iparomlimab Based Regimens for the Neoadjuvant Treatment of Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLIT-BTC
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tuvonralimab/Iparomlimab combination (Experimental)
  Interventions: Drug: Tuvonralimab/Iparomlimab combination with GEMOX chemotherapy

INTERVENTIONS:
Drug: Tuvonralimab/Iparomlimab combination with GEMOX chemotherapy — Tuvonralimab/Iparomlimab combination with GEMOX chemotherapy

SUMMARY:
The goal of this clinical trial is to learn if Tuvonralimab/Iparomlimab-based neoadjuvant regimens can improve surgical and pathological outcomes in adults (≥18 years) with resectable or borderline-resectable biliary tract cancer (intrahepatic/extrahepatic cholangiocarcinoma or gallbladder cancer), ECOG 0-1, and no prior neoadjuvant therapy.

The main questions it aims to answer are:

1. Does the regimen increase the R0 resection rate (negative margins)?
2. Does it raise major or pathologic complete response rates (MPR/pCR) and improve event-free survival (EFS) without increasing perioperative complications?

Researchers will compare Tuvonralimab/Iparomlimab-based therapy + GEMOX chemotherapy to surgery to see if immunotherapy leads to higher R0 resection, deeper pathologic response, and better EFS/PFS/OS with acceptable safety.

Participants will:

Undergo baseline assessments: imaging (contrast-enhanced CT/MRI ± PET), labs, histology, and optional biomarker sampling.

Receive neoadjuvant therapy: 2-4 cycles (\~6-12 weeks) of a Tuvonralimab/Iparomlimab-based regimen per protocol.

Have restaging by RECIST 1.1; eligible participants proceed to curative-intent surgery with central review of margins and tumor regression grading (TRG/MPR/pCR).

Receive protocol-directed postoperative management and safety monitoring (CTCAE v5.0) and be followed every 8-12 weeks for EFS, PFS, OS, conversion-to-resection rate, nodal down-staging, perioperative complications, length of stay, and any surgery delays.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and agreed to sign the written informed consent. They had good compliance and cooperated well with the follow-up.
* At the time of signing the informed consent form, the applicant was over 18 years old and could be of any gender.
* Patients with bile duct cancer diagnosed by histological or imaging methods, and whose imaging assessment or clinical assessment indicates borderline resectability
* There is at least one measurable lesion (as per the RECIST 1.1 criteria, this measurable lesion must have a spiral CT scan diameter of ≥ 10mm or the short diameter of a swollen lymph node of ≥ 15mm)
* Patient has not received any systematic treatment in the past
* The patient has locally advanced disease but no distant metastasis. Theoretically, a R0 resection can be achieved through complex resection combined with vascular reconstruction, but the risk is high.
* One of the following situations exists: 1. The main portal vein or a long segment of the hepatic artery on one side is affected, while the other side is still capable of supplying blood or draining. Vascular angioplasty or reconstruction can be performed. 2. The tumor involves the bile duct area beyond one secondary branch, but does not affect the primary branch on the opposite side. It is expected that the available residual liver and bile duct drainage can still be retained. 3. There is suspected regional lymph node metastasis (at the hepatic hilum, abdominal cavity), but there is no distant lymph node or peritoneal implantation.
* The ECOG score was 0-1 within one week before enrollment.
* The hematology and organ functions are adequate. Based on the laboratory test results obtained within 14 days prior to the start of the treatment (unless otherwise specified): Blood routine examination: (No blood transfusion, no use of G-CSF, no use of drugs for correction within 14 days before screening): Hb ≥ 90 g/L; Neutrophils ≥ 1.5 × 109/L; PLT ≥ 100 × 109/L. Biochemical examination: (No albumin transfusion within 14 days): Appropriate liver function: ALT and AST ≤ 2.5 × ULN; Bilirubin ≤ 2.0 × upper limit of normal; Appropriate renal function: Creatinine ≤ 1.5 × ULN, or creatinine clearance rate (CCr) > 50 mL/min (using the standard Cockcroft-Gault formula)
* Fertile women: Agree to abstain from sexual intercourse (avoiding heterosexual intercourse) during the treatment period and for at least 6 months after the last administration (or use a contraceptive method with a failure rate of less than 1% for contraception)
* Men agree to abstain from sexual intercourse (not having sex with the opposite sex) or to use contraceptive measures, and agree not to donate sperm.

Exclusion Criteria:

* Has previously received any systemic treatment
* ECOG score > 1 point
* It is confirmed that there is liver metastasis outside the liver.
* Pregnant women (with a positive pregnancy test before taking the medicine) or lactating women
* Those who are known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs, CTLA-4 monoclonal antibody drugs, or their components (or any excipients) are not eligible.
* Having undergone major surgical procedures (except for biopsy) within 4 weeks prior to the first drug treatment, or having an incomplete healing of the surgical incision
* Significant clinical cardiovascular and cerebrovascular diseases, including but not limited to acute myocardial infarction occurring within 6 months prior to enrollment, severe/unstable angina pectoris, cerebrovascular accident or transient cerebral ischemic attack, congestive heart failure (NYHA classification ≥ 2 grade); arrhythmias requiring anti-arrhythmic drug treatment (except for beta-blockers or digoxin); repeated electrocardiogram QTc interval > 480 milliseconds (ms)
* Impaired liver and kidney functions, including conditions such as jaundice, ascites, and/or bilirubin levels > 3×ULN, creatinine ratio > 3.5g/24 hours, or renal failure requiring blood or peritoneal dialysis. And/or urine routine shows urine protein ≥ ++ or confirmed 24-hour urine protein quantification > 1.0g
* There is a persistent infection of grade 2 or above (according to CTCAE version 5.0)
* Having a history of thromboembolic events within the past 6 months (including stroke and/or transient ischemic attack)
* Hypertension that has not been well controlled by antihypertensive drugs (systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg)
* Participants who have had active autoimmune diseases or autoimmune disease history in the past two years; those who have active, known, or suspected autoimmune diseases that may affect important organ functions or who already/possibly require systemic immunosuppressive therapy.
* Known active central nervous system (CNS) metastasis and/or cancerous meningitis
* Be prepared or have previously undergone organ or allogeneic bone marrow transplantation
* A known history of active tuberculosis (with the tuberculosis bacteria)
* Having a history of gastrointestinal bleeding within the past 6 months or having a clear tendency towards gastrointestinal bleeding, and having either a CTCAE 5.0 grade 3 or above gastrointestinal fistula or non-gastrointestinal fistula in the past or currently
* Known history of human immunodeficiency virus (HIV) infection
* Those with positive results for active hepatitis B or hepatitis C and who have not received regular treatment. During the screening period, HBV DNA must be ≥ 2000 IU/ml (or ≥ 104 copies/ml). They can be enrolled only after reducing it to < 2000 IU/ml (or < 104 copies/ml) using entecavir; for the enrolled subjects with Anti-HBc(+)/HBsAg (+)/HBV DNA < 2000 IU/ml or Anti-HBc(+)/HBsAg (-)/HBV DNA < 2000 IU/ml, they must receive antiviral treatment during the trial, which can be with the previously used drugs or entecavir or tenofovir.
* Severe non-healing wounds, ulcers or fractures
* There is drug abuse; or any medical, psychological or social condition that may affect the research, the patient's compliance, be unstable, or even potentially endanger the patient's safety.
* There are unresolved toxicities of grade >1 that were caused by any previous treatment/operation (CTCAE 5.0, except for hair loss, anemia, and hypothyroidism)
* Patients who have objective evidence of severe lung function impairment in the past and at present, such as a history of severe pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, or drug-related pneumonia
* Received potent CYP3A4 inhibitor treatment within 7 days prior to the study, or received potent CYP3A4 inducer treatment within 12 days prior to the study
* With other malignant tumors, but having had (within the past 5 years) or concurrently having other untreated malignant tumors, for cured skin basal cell carcinoma, skin squamous cell carcinoma, in situ breast cancer and in situ cervical cancer, treated superficial bladder cancer and prostate adenocarcinoma that underwent surgical treatment and whose PSA tumor marker was within the normal range
* After the researchers' comprehensive assessment of the patient's condition, it was determined that the patient was not suitable for participating in this study.
* At the same time, he/she is also participating in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | Baseline (≤28 days before first dose); Neoadjuvant completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng Bi et al. First-line iparomlimab and tuvonralimab (QL1706) or iparomlimab (QL1604) + bevacizumab (BEV) for unresectable hepatocellular carcinoma (HCC): Updated results from the phase Ib/II DUBHE-H-106 study.. JCO 43, 579-579(2025).
- [Result] Pierot L, Flandroy P, Turjman F, Berge J, Vallee JN, Bonafe A, Bracard S. Selective endovascular treatment of intracranial aneurysms using micrus microcoils: preliminary results in a series of 78 patients. J Neuroradiol. 2002 Jun;29(2):114-21. PMID 12297733